CLINICAL TRIAL: NCT00811642
Title: A Multicenter, Open Label Study to Evaluate Safety and Efficacy of Posaconazole Oral Suspension in Treatment of Invasive Fungal Infection
Brief Title: Posaconazole Treatment of Invasive Fungal Infection (IFI) (P05551)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05551
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Fungal Infection
Keywords: refractory or first line medication intolerable invasive fungal infection
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole (Experimental): Posaconazole 400 mg twice a day (BID) oral suspension for 12 weeks
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — 400mg BID oral suspension for 12 weeks
  Other Names: Noxafil

SUMMARY:
The purpose of this multicenter, open label study, is to evaluate the safety and efficacy of a 12-week treatment with Posaconazole Oral Suspension in participants with IFI

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-70 years male or female
* Identified or clinically diagnosed IFI participants or high risk population who are resistant to, or recurrent from, or intolerable to, or may suffer toxic reaction from standard antifungal treatment.
* Sign informed consent form

Exclusion Criteria:

* Female participants who are pregnant or are nursing.
* Participants with known or suspected hypersensitivity or idiosyncratic reaction to azole agents or amphotericin B
* Participants with progressive nervous system diseases( excluding those IFI caused)
* Participants who take the following drugs known with interference with azole antifungal preparations

  * terfenadine, cisapride, and ebastine within 24 hours before entry
  * astemizole at entry or within 10 days before entry
  * cimetidine, rifampin, carbamazepine, phenytoin, rifabutin, barbiturates, isoniazid atharanthine and anthracyclines within 24 hours before entry
* The drugs listed above are prohibited during the investigation
* Serious organ diseases except hematological disorder such as cardiac or neurologic disorders or impairment expected to be unstable or progressive during the course of this study (eg, seizures or demyelinating syndromes, acute myocardial infarction within 3 months of study entry, myocardial ischemia, congestive heart failure, atrial fibrillation with ventricular rate <60/min, or history of torsades de pointes, symptomatic ventricular or sustained arrhythmias), unstable electrolyte abnormalities.
* Participants having an ECG with a prolonged QTc interval: QTc greater than 450 msec for men and greater than 470 msec for women.
* Expected to take during investigation or is taking systemic antifungal treatment
* Participants with severe renal insufficiency (estimated creatinine clearance less than 50 mL/minute or likely to require dialysis during the study), ALT,AST AKP or total bilirubin are >2×ULN.
* Participants expected to survive no more than 72hrs
* Participants receiving artificial aeration and will not withdraw within 24hrs
* Participants who have used any investigational drugs or biologic agents or anticipated other clinical trials within 30 days of study entry.
* Prior enrollment in this study.
* History of alcohol and/or drug abuse.
* Participants cannot be compliant in investigator's opinion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Huang X, Wang F, Chen Y, Liu T, Wang J, Hu J, Jie J, Chen F, Wang S, Shen Z, Yu L, Yu K, Liang Y. A multicenter, open-label study of posaconazole oral suspension in the treatment of invasive fungal infections in patients refractory to or intolerant of first-line therapy. Future Microbiol. 2012 Feb;7(2):201-9. doi: 10.2217/fmb.11.158. PMID 22324990

RESULTS

PARTICIPANT FLOW:
Groups:
- Posaconazole: 400 mg twice a day (BID) oral suspension for
  12 weeks
Period: Overall Study
Arm/Group | Posaconazole
Started | 62 (63 participants were screened and enrolled; 62 participants from Safety Set (SS) started study drug.)
Completed | 47 (The Per Protocol Set (PPS) includes the 47 participants who completed the study per protocol.)
Not Completed | 15
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 7
Not completed — Cumulative use of antifungal agent | 2

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.41 (14.752)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 28
Region of Enrollment [Number; unit: participants]
  China | 62

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Had Clinical Response at 4 Weeks With Posaconazole Treatment
Description: EVALUATION OF PARTICIPANTS' CLINICAL RESPONSE BASED ON CRITERIA:
  Complete Response: resolution of IFI attributable symptoms, signs and laboratory or etiological abnormalities, if present at enrollment.
  Partial Response: clinically significant improvement in IFI attributable symptoms, signs and laboratory or etiological abnormalities, if present at enrollment, of which, one still had not achieved complete recession.
  Stable disease: no progress in IFI attributable symptoms, if present at enrollment.
  Failure: deterioration in IFI attributable clinical symptoms.
Time Frame: Treatment week 4
Population: Pool of participants were from the FAS: included all randomized participants who received at least one dose of study drug and who had valid data of primary efficacy endpoint for at least one follow-up visit after treatment. Did not include the 3 participants from the SS population (n=62) who withdrew from the study.
Measure: Number; unit: Particpants
Arm/Group | Posaconazole
Number analyzed (Participants) | 59
Particpants
  Complete response | 2 [52.88 to 80.9]
  Partial response | 39
  Stable disease | 11
  Failure | 7

2. Secondary Outcome: Number of Participants Who Had Clinical Response at 8 Weeks With Posaconazole Treatment
Description: as for outcome 1
Time Frame: Treatment week 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 59
Participants
  Complete response | 3 [46.38 to 75.4]
  Partial response | 34
  Stable disease | 11
  Failure | 11

3. Secondary Outcome: Number of Participants With Pathogenic Fungal Eradication at 4 Weeks With Posaconazole Treatment
Description: EVALUATION OF FUNGAL ERADICATION:
  Participants' mycological response to therapy was assessed by the following:
  Eradication: Negative culture or histologically documented absence of infecting
  fungal pathogen from a primary site previously positive.
  Presumed Eradication: Resolution of all IFI attributable symptoms, signs and laboratory or radiological abnormalities in which a repeat culture/biopsy was contraindicated.
  Persistence: Continued isolation of fungal pathogen from a primary site previously positive or cytological documentation of presence of fungal pathogen.
Time Frame: Treatment week 4
Population: Only FAS participants with positive fungal culture (of suspected site or blood) were evaluated. Last Observation Carried Forward (LOCF) was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 17
Participants
  Eradication | 2 [16.75 to 76.6]
  Presumed eradication | 6
  Disease persistence | 9

4. Secondary Outcome: Number of Participants With Pathogenic Fungal Eradication at 8 Weeks With Posaconazole Treatment
Description: as for outcome 3
Time Frame: Treatment week 8
Population: Only FAS participants with positive fungal culture (of suspected site or blood) were evaluated. LOCF was used for missing data.
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 17
Participants
  Eradication | 2 [16.75 to 76.6]
  Presumable eradication | 6
  Disease persistence | 9

5. Secondary Outcome: Number of Participants With Pathogenic Fungal Eradication at 12 Weeks With Posaconazole Treatment
Description: as for outcome 3
Time Frame: Treatment week 12
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 17
Participants
  Eradication | 2 [23.38 to 83.2]
  Presumable eradication | 7
  Disease persistent | 8

6. Secondary Outcome: Number of Participant Survivors at Week 14 of Post-Posaconazole Treatment Follow-up
Description: Total number of participant deaths was assessed at the end of 2 week post-treatment follow-up (14 weeks). The total number of deaths was compared to the number of survivors at baseline.
Time Frame: Follow-up week 14
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 59
Participants
  Survival | 57 [85.46 to 99.48]
  Death | 2

7. Primary Outcome: Number of Participants Who Had Clinical Response at 12 Weeks With Posaconazole Treatment
Description: EVALUATION OF PARTICIPANTS' CLINICAL RESPONSE BASED ON CRITERIA:
  Complete Response: resolution of Invasive Fungal Infection (IFI) attributable symptoms, signs and laboratory or etiological abnormalities, if present at enrollment.
  Partial Response: clinically significant improvement in IFI attributable symptoms, signs and laboratory or etiological abnormalities, if present at enrollment, of which, one still had not achieved complete recession.
  Stable disease: no progress in IFI attributable symptoms, if present at enrollment.
  Failure: deterioration in IFI attributable clinical symptoms.
Time Frame: Treatment week 12
Population: Pool of participants were from the Full Analysis Set (FAS): included all randomized participants who received at least one dose of study drug and who had valid data of primary efficacy endpoint for at least one follow-up visit after treatment. Did not include the 3 participants from the SS population (n=62) who withdrew from the study.
Measure: Number; unit: Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 59
Participants
  Complete response | 6
  Partial response | 32
  Stable | 11
  Failure | 10

ADVERSE EVENTS:
Description: 63 participants were screened and enrolled; 62 participants started on study drug and comprised the Safety Set (SS). SS population included randomized subjects who received at least one dose of study drug and valid data of safety endpoints was available for at least one follow-up visit after treatment.
Groups:
- POSACONAZOLE: 400mg oral suspension BID for 12 weeks
Arm/Group | POSACONAZOLE
Serious Adverse Events (participants affected / at risk) | 5/62
Other Adverse Events (participants affected / at risk) | 40/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POSACONAZOLE (N=62)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (2)
LUNG INFECTION (Infections and infestations) | 1 (1)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POSACONAZOLE (N=62)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 11 (12)
NAUSEA (Gastrointestinal disorders) | 9 (11)
VOMITING (Gastrointestinal disorders) | 4 (4)
FATIGUE (General disorders) | 5 (8)
OEDEMA PERIPHERAL (General disorders) | 7 (10)
PYREXIA (General disorders) | 14 (21)
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 6 (7)
LUNG INFECTION (Infections and infestations) | 5 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 16 (22)
HEADACHE (Nervous system disorders) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (6)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) agrees not to publish or publicly present any interim results of the Protocol study without the prior written consent of the Sponsor. PI further agrees to provide to the Sponsor thirty (30) days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the Protocol study. The sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts.